CLINICAL TRIAL: NCT06766825
Title: Phase II Proof-of-concept, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Plitidepsin in Adults with Post-COVID-19 Condition (PCC)
Brief Title: Study to Evaluate the Efficacy and Safety of Plitidepsin in Adults with Post-COVID-19 Condition (PCC)
Acronym: THALASSA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Collaborators: PharmaMar (Industry); IrsiCaixa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: THALASSA 2.0; 2024-516378-31-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-31; First posted 2025-01-09 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Post COVID-19 Condition; Long COVID Syndrome; Persistent COVID-19; Persistent COVID Condition; Long COVID
Keywords: SARS-CoV-2; COVID-19; Long COVID19; Plitidepsin
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19 | interventions — plitidepsin

STUDY DESIGN:
Intervention Model Description: Randomized (1:1:1), placebo-controlled, double-blind clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Masking of investigational products will ensure that both the investigator and the participant are blinded to the product administered. The pharmacist service will be responsible for masking the study treatments. Both treatments (Plitidepsin and placebo) have the same route of administration. All the participants (from all arms) will receive the pre-medication required for the plitidepsin treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- A. Plitidepsin Arm (Experimental): Subjects in arm A will receive the plitidepsin 1.5 mg/day 1h-IV during the four treatment periods on Days 1 to 3, Days 15 to 17, Days 29 to 31 and Days 43 to 45.
  Interventions: Drug: Plitidepsin 1.5 mg/day
- B. Placebo/Plitidepsin (Experimental): Subjects in arm B will receive 1h-IV placebo 1 vial /day during the first two treatment periods (Days 1 to 3 and Days 15 to 17) and plitidepsin 1.5 mg/day 1h-IV during the last two treatment periods (Days 29 to 31 and Days 43 to 45).
  Interventions: Drug: Placebo and Plitidepsin 1.5mg/day
- C. Placebo Arm (Placebo Comparator): Subjects in arm C will receive 1h-IV placebo 1 vial/day during the four treatment periods on Days 1 to 3, Days 15 to 17, Days 29 to 31, and Days 43 to 45.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Plitidepsin 1.5 mg/day — Receive 1.5 mg/day of plitidepsin intravenously (IV) over a 1-hour infusion for 3 consecutive days every 15 days during 4 treatment periods.
  The participant will receive the following pre-medication before receiving the study treatment:
  * Palonosetron 0.25 mg IV
  * Dexchlorpheniramine maleate 5 mg IV (or equivalent to H1 receptor antihistamines)
  * Famotidine 40 mg oral (60 minutes before starting the plitidepsin/placebo infusion)
  * Dexamethasone phosphate 8 mg IV (equivalent to 6.6 mg of dexamethasone)
  Premedication should be completed 20-30 minutes before starting the plitidepsin/placebo infusion.
  Arms: A. Plitidepsin Arm
Drug: Placebo — Receive placebo intravenously (IV) over a 1-hour infusion for 3 consecutive days every 15 days during 4 treatment periods.
  The participant will receive the following pre-medication before receiving the study treatment:
  * Palonosetron 0.25 mg IV
  * Dexchlorpheniramine maleate 5 mg IV (or equivalent to H1 receptor antihistamines)
  * Famotidine 40 mg oral (60 minutes before starting the plitidepsin/placebo infusion)
  * Dexamethasone phosphate 8 mg IV (equivalent to 6.6 mg of dexamethasone)
  Premedication should be completed 20-30 minutes before starting the plitidepsin/placebo infusion.
  Arms: C. Placebo Arm
Drug: Placebo and Plitidepsin 1.5mg/day — Receive placebo intravenously (IV) over a 1-hour infusion for 3 consecutive days every 15 days during two treatment periods and receive plitidepsin 1.5mg/day during the last two treatment periods.
  The participant will receive the following pre-medication before receiving the study treatment:
  * Palonosetron 0.25 mg IV
  * Dexchlorpheniramine maleate 5 mg IV (or equivalent to H1 receptor antihistamines)
  * Famotidine 40 mg oral (60 minutes before starting the plitidepsin/placebo infusion)
  * Dexamethasone phosphate 8 mg IV (equivalent to 6.6 mg of dexamethasone)
  Premedication should be completed 20-30 minutes before starting the plitidepsin/placebo infusion.
  Arms: B. Placebo/Plitidepsin

SUMMARY:
The study aims to prove that plitidepsin could be an efficacious, safe, and well-tolerated therapy for PCC. To this end, we will perform a randomized, double-blind study comparing the clinical and laboratory benefits of plitidepsin vs. placebo in 90 subjects with moderate to severe functional disability. The study consists of an intervention period and a follow-up period, with a total of 135 +/-3 days approximately between both periods.

During the intervention period, four treatment cycles will be administered, scheduled every 15 days (every 2 weeks), with intravenous (IV) infusion over three consecutive days. After completing the intervention period, a 90-day (+/-5) follow-up period will be conducted.

Subjects in arm A will receive the plitidepsin 1.5 mg/day 1h-IV during the four treatment periods on Days 1 to 3, Days 15 to 17, Days 29 to 31 and Days 43 to 45. Subjects in arm B will receive 1h-IV placebo 1 vial /day during the first two treatment periods and will receive the plitidepsin 1.5 mg/day 1h-IV during the last two treatment periods. Subjects in arm C will receive 1h-IV placebo 1 vial/day during the four treatment periods.

DETAILED DESCRIPTION:
Plitidepsin, a marine-derived cyclic depsipeptide that inhibits SARS-CoV-2 replication at nanomolar concentrations by targeting the host protein eukaryotic translation elongation factor 1A, could be a suitable candidate treatment for "Long COVID" because of a triple mechanism of action; a) it has demonstrated potent anti-SARS-CoV-2 in vitro activity, (b) it has a systemic anti-inflammatory effect, detailed in the text below, and (c) has an anti-herpes antiviral effect, which could provide additional therapeutic benefits to prevent herpesvirus reactivation seen in Long-COVID.

An interim analysis will be conducted upon reaching 30% and 50% of recruitment (patients treated with at least one dose and 28 days (+/- 2 days) of FUP)). The first interim analysis will focus exclusively on safety assessment, based on adverse events reported to date. The second interim analysis (50%) will evaluate safety and futility. A blinded safety report will be prepared, summarizing adverse events, and submitted to the Data Safety Monitoring Board (DSMB) for review and to determine whether to continue, modify, or terminate the study

ELIGIBILITY:
1. Male or female individuals 18 years old or older.
2. Evidence of SARS-CoV-2 infection at least 90 days prior to study recruitment, defined by either (a) nasopharyngeal SARS-CoV-2 nucleic acid test [polymerase chain reaction (PCR) or transcription mediated amplification (TMA)], (b) validated Nasopharyngeal Lateral Flow Assay rapid antigen test (RAT), or (c) or positive serology against SARS-CoV-2 N protein regardless vaccination status.
3. 3 or more symptoms of PCC affecting at least two organs, after 90 days from the onset of SARS-CoV2 infection and that last for at least 2 months and cannot be explained by an alternative diagnosis. Symptoms may be new onset following initial recovery from an acute COVID-19 episode or persist from the initial illness. Symptoms may also fluctuate or relapse over time.
4. Unable to perform all usual duties/activities, defined as grades 3 or 4 in PCFS (Annex 3).
5. Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study.
6. Having understood the information provided and capable of providing informed consent

EXCLUSION CRITERIA

1. Last SARS-CoV-2 vaccine dose during the previous 30 days.
2. Patients with active uncontrolled infections.
3. Patients infected by SARS-CoV-2 virus in the last 90 days prior to the screening visit.
4. Patients receiving treatment with strong cytochrome P450 3A4 (CYP3A4) inhibitors or inducers (Annex 1) throughout plitidepsin treatment period and until 24-h washout period.
5. Pacients receiving chronic glucocorticoid therapy (high-dose corticosteroids [ie, 20 mg of prednisone daily or equivalent for ≥2 weeks)
6. Any of the following cardiac conditions or risk factors:

   * Cardiac infarction or cardiac surgery episode within the last six months 14
   * History of known congenital QT prolongation;
   * Known structural cardiomyopathy with abnormal left ventricular ejection fraction (LVEF) <50%;
   * Current clinical evidence of heart failure or acute cardiac ischaemia (New York Heart Association (NYHA) class III-IV).
7. Hypersensitivity to the active ingredient or any of the excipients (mannitol, macrogolglycerol hydroxystearate, and ethanol) or contraindication to receive systemic glucocorticoids, antihistamine H1/H2 receptor agents, or antiserotonine 5HT3 receptors drugs.
8. Mast cell activation syndrome.
9. Females who are pregnant (negative serum or urine pregnancy test required for all females of childbearing potential at screening) or breast-feeding.
10. Females of childbearing potential (females who are not surgically sterile or postmenopausal defined as amenorrhea for >12 months) who are not using highly effective contraceptive methods, while on study treatment and for 6 months after last dose of plitidepsin. Fertile males with partners of childbearing potential must use condom during treatment and for 6 months after last dose of plitidepsin. Refer to Annex 2 for contraception requirements.
11. Unable to consent and/or comply with study requirements, in the opinion of the investigator.
12. Currently participating or participated in a clinical trial within the prior

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in the overall health in patients from each group using patient reported outcomes measurement information system score (PROMIS-29®). | On day 90 of follow-up period
  Difference between groups on the patient-reported outcomes measurement information system (PROMIS-29®) score health scale measured by T-Score; Each domain is scored on a 5-point scale, (without any difficulty, with a little difficulty, with some difficulty, with much difficulty, unable to do), in case of the pain domain is on a 10-point scale; from no pain to the worse pain. on day 90 (±5) of the follow-up period* (after the intervention).

SECONDARY OUTCOMES:
To compare the safety/tolerability of Plitidepsin Vs placebo in terms of adverse events in patients with PCC. | On day 90 of follow-up period
  The proportion of adverse events (AE, coded by MedDRA) comparing between groups at day 90 (±5) of the follow-up period, considering:
  1. All AEs.
  2. AEs grade 3 and 4 leading to discontinuation from the study.
  3. AEs of special interest (AESI): cardiac, liver, acute-infusional reactions.
To compare the incidence of Treatment-Emergent Adverse Events (TEAEs) between groups. | On day 10, day 30 and day 90 of follow-up period
  Percentage of TEAEs detected on day 10 (±2), day 30 (±2), and day 90 (±5) of the follow-up period.
To compare changes in the overall health in patients from each group using patient reported outcomes measurement information system score (PROMIS-29®). | On day 10, day 30 and day 90 of follow-up period
  Difference between groups on the PROMIS-29® health scale measured by T-Score on day 10 (±2), day 30 (±2), and day 90 (±5) of the follow-up period. Each domain is scored on a 5-point scale, (without any difficulty, with a little difficulty, with some difficulty, with much difficulty, unable to do), in case of the pain domain is on a 10-point scale; from no pain to the worse pain. on day 90 (±5) of the follow-up period* (after the intervention).
To compare functional capacity changes in patients from each group using the post-COVID-19 Functional State (PCFS) scale. | On day 10, day 30 and day 90 of follow-up period
  Difference between groups in functional capacity on the PCFS scale on day 10 (±2), day 30 (±2), and day 90 (±5) of the follow-up period.
To compare symptomatic changes in patients from each group using the Can Ruti Questionnaire. | On day 10, day 30 and day 90 of follow-up period
  Proportion of subjects with ≥10 points reduction in the Can Ruti Questionnaire scale on day 10 (±2), day 30 (±2), and day 90 (±5) of the follow-up period.
To compare changes in terms of Quality of Life (QoL) for each group. | On day 10, day 30 and day 90 of follow-up period
  Difference between groups according to the EuroQoL-5D questionnaire on day 10 (±2), day 30 (±2), and day 90 (±5) of the follow-up period.
To compare neuropsychological symptomatology [psychomotor speed and executive function] in patients with PCC among the three treatment arms. | On day 10, day 30 and day 90 of follow-up period
  Change from baseline** in neuropsychological symptoms to day 10 (±2), day 30 (±2), and day 90 (±5) of the follow-up period, measured using NeuScreen questionnaire to evaluate the psychomotor speed and executive function measured in seconds.
To compare neuropsychological symptomatology [depressive symptoms] in patients with PCC among the three treatment arms. | On day 10, day 30 and day 90 of follow-up period
  Change from baseline** in neuropsychological symptoms to day 10 (±2), day 30 (±2), and day 90 (±5) of the follow-up period, using the PHQ-9 score questionnaire to evaluate the depressive symptoms, each question is scored on a 4-point scale, where (0) is the most positive answe and (3) is the worse condition.
To compare neuropsychological symptomatology [ anxiety symptoms] in patients with PCC among the three treatment arms. | On day 10, day 30 and day 90 of follow-up period
  Change from baseline** in neuropsychological symptoms to day 10 (±2), day 30 (±2), and day 90 (±5) of the follow-up period, using the GAD-7 questionnaire to evaluate anxiety symptoms; Each question is scored as follows: 0 points: "Not at all", 1 point: "Several days", 2 points: "More than half the days", 3 points: "Nearly every day"
To compare neuropsychological symptomatology [sleep quality] in patients with PCC among the three treatment arms. | On day 10, day 30 and day 90 of follow-up period
  Change from baseline** in neuropsychological symptoms to day 10 (±2), day 30 (±2), and day 90 (±5) of the follow-up period, measured using PSQI to evaluate sleep quality; the scores for the seven components are then summed to yield a global PSQI score, which ranges from 0 to 21. A global score greater than 5 suggests poor sleep quality.
To compare neuropsychological symptomatology [disability] in patients with PCC among the three treatment arms. | On day 10, day 30 and day 90 of follow-up period
  Change from baseline** in neuropsychological symptoms to day 10 (±2), day 30 (±2), and day 90 (±5) of the follow-up period, using WHODAS 2.0 questionnaire to evaluate disability: Each item is scored on a scale from 1 to 5, with higher scores indicating greater difficulty in functioning. The total score is calculated by summing the scores for all items, and it can be converted into a standardized score ranging from 0 to 100, where higher scores indicate greater disability.
To compare changes in terms of physical activity in patients with PCC among the three arms. | On day 10, day 30 and day 90 of follow-up period
  Change from baseline in physical activity to day 10 (±2), day 30 (±2), and day 90 (±5) of the follow-up period, assessed using the International Physical Activity Questionnaire (IPAQ).
To compare changes in terms of fatigue (Fatigue scale) in patients with PCC among the three treatment arms. | On day 10, day 30 and day 90 of follow-up period
  Change from baseline in physical activity to day 10 (±2), day 30 (±2), and day 90 (±5) of the follow-up period, evaluated using the Fatigue Severity Scale (FSS): nine statements, of 7-point Likert scale, where (1- Strongly disagree) and (7-Strongly agree). Higher scores indicate greater fatigue severity.
To compare changes in terms of fatigue (Five times sit to stant test) in patients with PCC among the three treatment arms. | On day 10, day 30 and day 90 of follow-up period
  Change from baseline in physical activity to day 10 (±2), day 30 (±2), and day 90 (±5) of the follow-up period, evaluated using Five Times Sit-to-Stand Test (5xSTS), The score is the total time in seconds
To compare the evolution of inflammation markers in patients with PCC among the three arms. | On day 10, day 30 and day 90 of follow-up period
  Change from baseline in inflammation markers on day 10 (±2), day 30 (±2), and day 90 (±5) of the follow-up period.
To compare immune response markers: Antinuclear antibodies (ANAs) in patients with persistent COVID among the three treatment arms. | On day 10, day 30 and day 90 of follow-up period
  Change from baseline in Antinuclear antibodies (ANAs) to day 10 (±2), day 30 (±2), and day 90 (±5) of the follow-up period. measured in UI/mL.
To compare immune response markers: antiphospholipid antibodies (Abs) in patients with persistent COVID among the three treatment arms. | On day 10, day 30 and day 90 of follow-up period
  Change from baseline in antiphospholipid antibodies (Abs),) to day 10 (±2), day 30 (±2), and day 90 (±5) of the follow-up period. measured in UI/mL.
To compare immune response markers: antimitochondrial antibodies in patients with persistent COVID among the three treatment arms. | On day 10, day 30 and day 90 of follow-up period
  Change from baseline in antimitochondrial antibodies to day 10 (±2), day 30 (±2), and day 90 (±5) of the follow-up period. measured in UI/mL.
To compare the SARS-CoV-2 RNA antigenemia (presence of viral components) in plasma with persistent COVID among the three treatment arms. | On day 10, day 30 and day 90 of follow-up period
  Change from baseline in viral components (SARS-CoV-2 RNA antigenemia) in plasma to day 10 (±2), day 30 (±2), and day 90 (±5) of the follow-up period. The SARS-CoV-2 RNA is quantified in pg/mL.
To compare alterations in Complement Activitation: Hemolytic Complement CH50 in patients with persistent COVID among the three treatment arms. | On day 10, day 30 and day 90 of follow-up period
  Change from baseline in Complement Activity: Hemolytic Complement CH50 to day 10 (±2), day 30 (±2), and day 90 (±5) of the follow-up period. measured in UI/mL.
To compare alterations in thromboinflammatory components (prothrombin time (PT)), among the three treatment arms. | On day 10, day 30 and day 90 of follow-up period
  Change from baseline in prothrombin time (PT) ratio in plasma to day 10 (±2), day 30 (±2), and day 90 (±5) of the follow-up period.
To compare alterations in thromboinflammatory components (activated partial thromboplastin time (aPTT)), among the three treatment arms. | On day 10, day 30 and day 90 of follow-up period
  Change from baseline in activated partial thromboplastin time (aPTT) in seconds, in plasma to day 10 (±2), day 30 (±2), and day 90 (±5) of the follow-up period.
To compare alterations in thromboinflammatory components (D-Dimer), among the three treatment arms. | On day 10, day 30 and day 90 of follow-up period
  Change from baseline in D-Dimer measured in ng/mL, in plasma to day 10 (±2), day 30 (±2), and day 90 (±5) of the follow-up period.
To compare alterations in thromboinflammatory components (Fibrinogen), among the three treatment arms. | On day 10, day 30 and day 90 of follow-up period
  Change from baseline in Fibrinogen measured in mg/dL, in plasma to day 10 (±2), day 30 (±2), and day 90 (±5) of the follow-up period.
To compare alterations in thromboinflammatory components (Antithrombin III (ATIII)), among the three treatment arms. | On day 10, day 30 and day 90 of follow-up period
  Change from baseline in Antithrombin III (ATIII) measured in %, in plasma to day 10 (±2), day 30 (±2), and day 90 (±5) of the follow-up period.
To compare alterations in thromboinflammatory components (Factor de Von willebrand), among the three treatment arms. | On day 10, day 30 and day 90 of follow-up period
  Change from baseline in Factor de Von Willebrand measured in %, in plasma to day 10 (±2), day 30 (±2), and day 90 (±5) of the follow-up period.
To compare alterations in hormonal components (Serotonin) among the three treatment arms. | On day 10, day 30 and day 90 of follow-up period
  Change from baseline in serotonin (UI) in plasma to day 10 (±2), day 30 (±2), and day 90 (±5) of the follow-up period.
To compare alterations in hormonal components (Dopamine) among the three treatment arms. | On day 10, day 30 and day 90 of follow-up period
  Change from baseline in dopamine alterations in plasma to day 10 (±2), day 30 (±2), and day 90 (±5) of the follow-up period. measured in ug/24 h

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No